CLINICAL TRIAL: NCT05800665
Title: A Phase 1, Open-Label, Multicenter, Dose-Escalation and Expansion Study Evaluating the Safety, Pharmacokinetics, and Activity of RO7656594 in Patients With Advanced or Metastatic Prostate Cancer
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Activity of RO7656594 In Participants With Advanced or Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO44537; 2023-504013-68-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Prostate Cancer; Metastatic Prostate Cancer
Keywords: Castration-resistant
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage 1: Dose Escalation (Experimental): Participants will receive RO7656594 administered at a specified dose on specific days in each 28-day cycle. The dose will be increased in successive cohorts until a study-specific threshold is reached.
  Interventions: Drug: RO7656594
- Stage 2: Expansion (Experimental): Participants will receive RO7656594 at or below the maximum tolerated dose (MTD) or maximum administered dose (MAD).
  Interventions: Drug: RO7656594

INTERVENTIONS:
Drug: RO7656594 — RO7656594 will be administered orally at specified dose on specified days.
  Other Names: GDC-2992

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and preliminary activity of RO7656594 in participants with advanced or metastatic prostate cancer. It will also identify recommended doses and regimens for RO7656594 for subsequent studies.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
2. Metastatic prostate adenocarcinoma without small-cell carcinoma or neuroendocrine features.
3. Prior therapy with a second-generation androgen receptor (AR)-targeted therapy (e.g., abiraterone, enzalutamide, apalutamide, darolutamide).
4. Prior therapy with a taxane regimen or are considered ineligible for treatment with a taxane regimen or have refused treatment with a taxane regimen, unless otherwise specified.
5. For participants with a known pathogenic breast cancer gene 1 (BRCA1) or BRCA2 mutation: prior therapy with a poly (adenosine diphosphate (ADP)-ribose) polymerase (PARP) inhibitor, or are considered ineligible for treatment with a PARP inhibitor, if such therapy is approved and available.

Key Exclusion Criteria:

1. Treatment with any approved systemic anti-cancer therapy within 14 days or 5 drug elimination half-lives (whichever is longer, not to exceed 28 days) prior to the first study treatment.
2. Treatment with any investigational agent within 28 days prior to the first study treatment.
3. Treatment with any previous AR protein degrader.
4. Untreated central nervous system (CNS) metastases or leptomeningeal disease.

Note: Other protocol specified inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | From Cycle 1 Day 1 until 28 days after the final dose (Up to approximately 24 months) (1 cycle= 28 days)
Percentage of Participants Who Experience Dose-limiting Toxicities (DLTs) | Days 1-28 of Cycle 1

SECONDARY OUTCOMES:
Plasma Concentration of RO7656594 | Multiple timepoints from Cycle 1 Day 1 up to approximately 12 months (1 cycle= 28 days)
  The pharmacokinetics (PK) of RO7656594 will be evaluated in plasma.
Prostate-Specific Antigen-30% (PSA30) Response Rate of RO7656594 | From Cycle 1 Day 1 until 28 days after the final dose (Up to approximately 24 months) (1 cycle= 28 days)
Prostate-Specific Antigen-50% (PSA50) Response Rate of RO7656594 | From Cycle 1 Day 1 until 28 days after the final dose (Up to approximately 24 months) (1 cycle= 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (25):
- United States (5):
  - HonorHealth, Scottsdale, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Sarah Cannon Research Institute @ Florida Cancer, Orlando, Florida
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - SCRI Oncology Partners, Nashville, Texas
- Australia (4):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Macquarie University Hospital, New South Wales, New South Wales
  - Monash Health Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
- Canada (2):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- France (2):
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
- Spain (4):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Clinica Universidad de Navarra-Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
- United Kingdom (4):
  - Cambridge Clinical Research Centre, Cambridge
  - Leicester Royal Infirmary, Leicester
  - The Christie, Manchester
  - Royal Marsden Hospital - Surrey, Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing